CLINICAL TRIAL: NCT03807817
Title: Synergistic Effects of Anxiety and Alcohol Use Among Latinos and Its Sociocultural Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Andres G. Viana, Assistant Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1K23AA025920-01A1 (NIH)
Record Dates: First submitted 2019-01-07; First posted 2019-01-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Alcohol Drinking; Racism
MeSH Terms: conditions — Alcohol Drinking; Racism | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Moderate Alcohol (Experimental)
  Interventions: Other: Alcohol administration
- Low Alcohol (Experimental)
  Interventions: Other: Alcohol administration
- Placebo Alcohol (Active Comparator)
  Interventions: Other: Placebo
- No Alcohol (Active Comparator)
  Interventions: Other: No Alcohol

INTERVENTIONS:
Other: Alcohol administration — Amount of alcohol to be administered.
  Arms: Low Alcohol; Moderate Alcohol
Other: Placebo — Placebo Alcohol
  Arms: Placebo Alcohol
Other: No Alcohol — No Alcohol
  Arms: No Alcohol

SUMMARY:
The purpose of this study is to examine the pharmacological effects of alcohol on acute anxiety levels in a sample of Latino drinkers, and cultural experiences influencing these relationships.

ELIGIBILITY:
Inclusion Criteria:

1. 21-65 years of age
2. moderate or heavy drinker based on a past-month AUDIT score >= 8.

Exclusion Criteria:

1. Possibility of being pregnant (verified by urine sample);
2. Self-reported history of or treatment for alcohol/other drug problems (as required by the IRB in past human alcohol administration research);
3. Moderate risk for drug problems as indicated by SMAST scores ≥ 5 or ASSIST scores of ≥ 4 (see Measures);
4. Medical conditions that contraindicate the use of alcohol (e.g., diabetes, liver disease);
5. Current use of psychiatric meds or any meds with alcohol contraindication (e.g., antibiotics);
6. Current non-alcohol substance use disorder;
7. Active suicidality (i.e., suicidal ideation, intent, and/or plan) or current psychosis.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory, State Version (STAI-S) | 5 minutes before alcohol administration, and 5 minutes after alcohol administration.
  The State-Trait Anxiety Inventory, State Version (STAI-S) is a 20-item self-report questionnaire which assesses state (i.e., current) anxiety. Participants are asked to rate the frequency with which they experience a variety of anxiety symptoms (e.g., "I feel nervous and restless") on a 4-point scale (1 = almost never to 4 = almost always). Total scores (range = 20-80) are computed by summing individual item scores; higher scores indicate higher state anxiety.
  The State-Trait Anxiety Inventory, State Version (STAI-S) will be used to measure manifest anxiety among participants 5 minutes before, and 5 minutes after, the alcohol administration. We will specifically measure changes in manifest anxiety from pre- to post-alcohol administration by subtracting the participant's score on the STAI-S after the alcohol administration from the participant's score on the STAI-S before the alcohol administration.
Alcohol Urge Questionnaire (AUQ) | 5 minutes before alcohol administration, and 5 minutes after alcohol administration.
  Urge to drink will be measured using the internally consistent, reliable, and well-validated Alcohol Urge Questionnaire (AUQ), an 8-item measure of state (current) urge to drink alcohol. Items are rated on a 7-point scale from 1 = "strongly disagree" to 7 = "strongly agree." A total score is computed by adding responses to each of the items. Higher scores indicate a stronger urge to drink.
  The Alcohol Urge Questionnaire (AUQ) will be used to measure urge to drink among participants at 5 minutes before, and 5 minutes after, the alcohol administration. We will specifically measure changes in urge to drink from pre- to post-alcohol administration by subtracting the participant's score on the AUQ post-alcohol administration from the participant's score on the AUQ pre-alcohol administration.
Amount of alcohol consumed in "standard drinks" (0.6 oz. ethanol equivalents, 12 oz. U.S. domestic beer, 5 oz. 12% alcohol table wine, 1.5 oz. 80-proof hard liquor) | 5 minutes after participating in the stressor task.
  Amount of alcohol consumed in "standard drinks" (0.6 oz. ethanol equivalents, 12 oz. U.S. domestic beer, 5 oz. 12% alcohol table wine, 1.5 oz. 80-proof hard liquor) will be estimated for each participant.

SECONDARY OUTCOMES:
Kulis, Marsiglia & Nieri's (2009) Substance Use Attitudes/Expectancies Scale | 5 minutes before alcohol administration.
  We will examine participants' Substance Use Attitudes and Expectancies 5 minutes before the intervention using Kulis, Marsiglia & Nieri's (2009) Substance Use Attitudes/Expectancies Scale. The scale contains 12 items, rated from 1 = "definitely no" to 4 = "definitely yes." Total scores are computed by averaging responses across items. Higher scores indicate more frequent pro-drug attitudes.

CONTACTS AND LOCATIONS:
Overall Officials: Andres G Viana, Ph.D., Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Data will be released directly by the investigators provided that those requesting the data can provide proof of their institution's IRB approval for planned analyses of the data. The investigator's team will be available to address queries.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available 2 years after completion of the study.
Access Criteria: We will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Data will be released directly by the investigators provided that those requesting the data can provide proof of their institution's IRB approval for planned analyses of the data.